CLINICAL TRIAL: NCT01477281
Title: A Clinical Multicenter, Phase III, Prospective, Randomized, Double-blind, Comparative Study to Evaluate the Efficacy and Tolerability of Venaflon Use in Reducing the Symptoms Caused by Chronic Venous Insufficiency When Compared With Daflon
Brief Title: Study to Evaluate the Efficacy and Tolerability of Venaflon Use in Reducing the Symptoms Caused by Chronic Venous Insufficiency When Compared With Daflon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório Teuto Brasileiro S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E01-TEU-VEN-08-10
Record Dates: First submitted 2011-10-19; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Venous Insufficiency; Disease
Keywords: chronic venous insufficiency; Daflon; Venaflon
MeSH Terms: conditions — Disease | interventions — Diosmin; Hesperidin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venafon (Diosmin and Hesperidin) (Experimental): Administer one tablet 2 times daily (oral), the main meals (lunch and dinner).
  Interventions: Drug: Daflon
- Daflon (Active Comparator): Administer one tablet 2 times daily (oral), the main meals (lunch and dinner).
  Interventions: Drug: Venaflon (Diosmin and Hesperidin)

INTERVENTIONS:
Drug: Daflon — Administer one tablet 2 times daily (oral), the main meals (lunch and dinner).
  Arms: Venafon (Diosmin and Hesperidin)
Drug: Venaflon (Diosmin and Hesperidin) — Administer one tablet 2 times daily (oral), the main meals (lunch and dinner).
  Arms: Daflon

SUMMARY:
The objective is to evaluate the effectiveness of the safety of Daflon in decreasing symptoms resulting from chronic venous insufficiency when compared with Daflon.

DETAILED DESCRIPTION:
"A clinical multicenter, phase III, prospective, randomized, double-blind, comparative study to evaluate the efficacy and tolerability of Venaflon use in reducing the symptoms caused by chronic venous insufficiency when compared with Daflon."

ELIGIBILITY:
Inclusion Criteria:

* Patients of any ethnic group, both sexes and aged at least 18 years and a maximum of 65 years
* Women and men of childbearing age who agree to use acceptable contraception throughout the study.
* Be patient with chronic venous insufficiency of lower limbs varicose comDiagnostico clinical CEAP 0-3 by CEAP
* Presence of at least 23 symptoms (pain, heaviness and discomfort, symptoms of heat and burning sensation in the legs) in the lower limbs, with a score equal to or greater than 4, as measured by visual analog scale
* Being the 7 days without any medication or treatment related to the venous system.
* Patients able to make proper use of medication
* Patients who consent to participate in the study by signing the Instrument of Consent.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Women who are breastfeeding
* Women and men of childbearing age who do not accept to use acceptable contraception throughout the study
* Patients under 18 or over 65 years
* Patients with a history of hypersensitivity to any component of the formula
* Presence of signs and symptoms of different conditions of venous disease to justify the pain or swelling
* Use of elastic compression in the last two weeks
* Venous obstruction of the lower limbs
* Patients who have previously used or Venaflon Daflon and did not benefit;
* Deep vein thrombosis in the last 6 months before entering the study;
* Use of diuretics in the last 4 weeks
* Previous venous surgery
* Patients with renal and liver failure
* Patients with gastritis or gastric ulcer
* Patients with blood clotting disorders
* Any condition which in the opinion of the physician researcher is significant and can make the patient unsuitable for study or you can place it under additional risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Improves the symptoms of chronic venous insufficiency with classification CEAP 0-3 | 30 days
  To evaluate the efficacy of Venaflon compared with Daflon in the improves of symptomatic treatment of chronic venous insufficiency with classification CEAP 0-3

SECONDARY OUTCOMES:
Identify adverse events, as well as their frequency and causality related to study medication. | 30 days
  The secondary outcome measure will be to evaluate the tolerability of Venaflon in the symptomatic treatment of chronic venous insufficiency with classification CEAP 0-3.